CLINICAL TRIAL: NCT00323219
Title: Oral Moxifloxacin Versus Cefazolin and Oral Probenecid in the Management of Skin and Soft Tissue Infections in the Emergency Department
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of British Columbia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PO3-0153
Record Dates: First submitted 2006-05-08; First posted 2006-05-09 (Estimated); Last update posted 2012-02-08 (Estimated); Status verified 2012-02

CONDITIONS: Cellulitis
Keywords: Cellulitis, RCT, emergency Department, Double-blind, Equivalence trial, Moxifloxacin, Cefazolin, Probenecid.
MeSH Terms: conditions — Cellulitis; Emergencies | interventions — Cefazolin; Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Cefazolin and Moxifloxacin — See Detailed Description.

SUMMARY:
Patients often come to the emergency department with bacterial skin infections (known as "cellulitis"). Some patients with very severe infections are admitted to hospital for antibiotic treatment and some are sent home on oral antibiotics. Many patients have moderate infections and are treated as outpatients with daily intravenous antibiotics for 2-5 days. In this patient group it is unclear if treatment with oral antibiotics is as effective as intravenous antibiotics. The purpose of this study is to determine if treatment of moderate cellulitis with an intravenous antibiotic (cefazolin) for 3-5 days is as effective as treatment with an oral antibiotic (moxifloxacin). We hypothesize that the oral agent will be as effective as intravenous treatment for moderate cellulitis.

DETAILED DESCRIPTION:
Extended description of the protocol, including information not already contained in other fields.

Objective: To compare 400 mg of oral moxifloxacin (Oral Group) once daily to 2 grams of IV cefazolin and 1 gram of oral probenecid once daily (IV group) for the treatment of moderate cellulitis.

Patients: Any patient presenting to the emergency department at St Paul's Hospital in Vancouver with a diagnosis of cellulitis requiring IV antibiotics, without contraindications to any of the study treatments, and not requiring hospital admission.

Assessments: Daily assessments are performed double-blind at 0, 1, 2, 3, 4, 5, 6, 7 and 14 days.

Primary outcome: Clinical cure at 7 days (resolution of symptoms, no change in antibiotic, no adverse events requiring discontinuation of study drug, no admission to hospital).

Secondary outcomes: Area of erythema, days of treatment, side-effects of medication, cost of treatment, patient satisfaction, relapse at 14 days.

Sample size: Based on equivalence of treatments a total of 390 patients are required (195/group).

ELIGIBILITY:
Inclusion Criteria:

* Cellulitis requiring outpatient intravenous antibiotic therapy;
* ability to understand,/sign informed consent;
* no contraindications to study medications,
* not pregnant/breastfeeding

Exclusion Criteria:

-

Max Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 390 (Estimated)
Dates: Start 2004-01; Primary Completion 2012-12 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Clinical cure at 7 days | 7 days

SECONDARY OUTCOMES:
Area of erythema (Days 0, 1, 2, 3, 4, 5, 6, 7), days of treatment, side-effects of medication, cost of treatment, patient satisfaction, relapse at 14 days | 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Rob Stenstrom, MD, Principal Investigator — The University of British Columbia
Locations (1):
- St. Paul's Hospital, Providence Healthcare, Emergency Medicine, Vancouver, British Columbia, Canada